CLINICAL TRIAL: NCT02985658
Title: Expanded Access Protocol With ABT-888 (Veliparib) in Patients With Metastatic BRCA-Mutation Associated or Triple Negative Breast Cancer
Brief Title: Expanded Access With ABT-888 (Veliparib) to Treat Metastatic Breast Cancer
Status: No longer available | Type: Expanded Access
Sponsor: University of Washington (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: 9763; RG1716061 (Other: Fred Hutch/University of Washington Cancer Consortium); NCI-2020-11567 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-12-05; First posted 2016-12-07 (Estimated); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Metastatic Breast Cancer With BRCA 1 or BRCA 2 Genetic Mutation; Triple-Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — veliparib; Cisplatin; Vinorelbine

INTERVENTIONS:
Drug: Veliparib — Patients will start veliparib at 300 mg po BID days 1 through 21 of the first 21 day cycle, then increase to 400 mg po BID days 1 through 21 of each subsequent cycle, as tolerated by the patient.
  At the treating investigator's discretion, and with principal investigator approval, veliparib may be used in combination with cisplatin and/or vinorelbine. Veliparib (300mg) will be dosed po BID on Days 1 through 14 of each 21-day cycle.
  The patient will receive therapy as long as there is therapeutic benefit
  Other Names: ABT-888
Drug: Cisplatin — Cisplatin will be administered intravenously (75 mg/m2) on Day 1 of each cycle
  Other Names: Platinol-AQ; Platinol
Drug: Vinorelbine — Vinorelbine will be administered intravenously on Day 1 and Day 8 of each 21-day cycle
  Other Names: Navelbine

SUMMARY:
This is an expanded access protocol to allow continued maintenance therapy with ABT-888 (veliparib) for three patients with metastatic triple negative breast cancer who are currently receiving the investigational product in association with clinical trial participation. Additionally, the protocol will enroll up to 7 new patients with metastatic BRCA associated or triple negative breast cancer to allow for additional access to veliparib monotherapy, or at the investigator's discretion, veliparib in combination with cisplatin and/or vinorelbine.

DETAILED DESCRIPTION:
ABT-888 (Veliparib) or Poly(ADP-ribose)-polymerase (PARP) is a nuclear enzyme that recognizes deoxyribonucleic acid (DNA) damage and facilitates DNA repair. Inactive PARPs 1 and 2 bind to damaged DNA, which leads to their auto-activation. The resulting activated PARP then poly(ADP-ribosyl)ates many nuclear target proteins, including those that facilitate DNA repair of both single-stranded or double-stranded DNA breaks. Thus, PARP inhibition will result in less efficient DNA repair following a DNA damage insult.

Since cancer cells are genetically unstable, often exhibiting complex karyotypes that include large deletions, insertions, and unbalanced translocations of chromosomal fragment, these cells are more susceptible than normal tissues to cytotoxicity induced by DNA-damaging agents.Of these, deficiencies in mismatch repair and homologous recombination are associated with the largest number of malignancies, including many sporadic TNBCs. These deficiencies render cells more dependent on PARP for DNA repair and, hence, are more prone to cytotoxicity induced by PARP inhibition. In particular, tumor cells with BRCA1 or BRCA2 deficiencies are exquisitely sensitive to PARP inhibition, even in the absence of any other insults. Identification of sporadic TNBC with defects in homologous recombination and mismatch repair independent of germline mutation of BRCA 1 and 2 is an active area of research interest.

PARP-enabled DNA repair may also compensate for the loss of other repair pathways. Higher expression of PARP in cancer cells compared to normal cells has been linked to drug resistance and the overall ability of cancer cells to sustain genotoxic stress.

The combination of platinum based chemotherapy and PARP inhibition may be most effective in TNBC, and particularly in subsets of TNBC. This combination may also be active in tumors with a germline BRCA1-deficiency and/or basal phenotype, since a defect in the DNA double-strand break repair pathway should increase sensitivity to these agents. The addition of a PARP inhibitor to platinum based chemotherapy may induce a "double hit" to tumor cells lacking homologous recombination without causing excess toxicity to normal cells. ABT-888 may be used in combination with the DNA damaging agent, cisplatin, to potentiate its cytotoxic effect and with vinorelbine to enhance tumor response rate. Safety and preliminary efficacy of veliparib in combination with cisplatin and vinorelbine in patients with advanced triple negative and BRCA-associated breast cancer has been reported.

ELIGIBILITY:
1. Inclusion Criteria Roll-over patients: This protocol allows for the inclusion of 3 patients actively participating in protocol 7161 who are expected to continue to benefit from uninterrupted dosing of veliparib monotherapy.

   For newly enrolled patients the following criteria should be satisfied within 28 days of Day 1 of protocol treatment. Results from routine clinical evaluations within 28 days prior to enrollment may be used to determine eligibility:
   * Locally recurrent and not amenable to surgical therapy, and/or metastatic breast cancer
   * Confirmed HER2-, BRCA1 or BRCA2 mutation-associated breast cancer or sporadic triple negative breast cancer.
   * No opportunity to receive veliparib under a current clinical trial.
   * Patients may have had any number of prior lines of chemotherapy, endocrine therapy, immunologic, or biologic regimens for metastatic breast cancer.
   * Patients receiving bisphosphonates, denosumab or LHRH-agonists are eligible.
   * 18 years and older.
   * Performance status > 60% on the Karnofsky scale (ECOG < 2).
   * Adequate hematologic, renal and hepatic function as follows:
   * Bone Marrow: Absolute neutrophil count (ANC) > 1,500/mm3 (1.5 × 109/L); Platelets > 100,000/mm3 (100 × 109/L); Hemoglobin > 9.0 g/dL
   * Serum creatinine < 1.5 × upper normal limit of institution's normal range OR creatinine clearance > 50 mL/min/1.73m2 for patients with creatinine levels above institutional normal;
   * Hepatic function: AST and/or ALT < 2.5 × the upper normal limit of institution's normal range.

     o For patients with liver metastases, AST and/or ALT < 5 × the upper normal limit of institution's normal range;
   * Bilirubin < 1.5 × the upper normal limit of institution's normal range;

     o Patients with Gilbert's Syndrome may have a bilirubin > 1.5 × the upper normal limit of institution's normal range.
   * Women of childbearing potential must agree to use adequate contraception (one of the following listed below) prior to protocol entry, for the duration of protocol participation and for 90 days following completion of therapy. Women of childbearing potential must have a negative serum pregnancy test within 21 days prior to initiation of treatment and/or be confirmed as having postmenopausal status. Criteria for determining menopause include any of the following: prior bilateral oopherectomy; age > 60 years; age < 60 years and amenorrheic for at least 12 months in the absence of chemotherapy, endocrine therapy, or ovarian suppression and FSH and estradiol in the postmenopausal range.
   * Total abstinence from sexual intercourse (minimum one complete menstrual cycle);
   * Vasectomized partner of female patients;
   * Hormonal contraceptives (oral, parenteral or transdermal) for at least 3 months prior to study drug administration;
   * Double-barrier method (condoms, contraceptive sponge, diaphragm or vaginal ring with spermicidal jellies or cream);
   * IUD (Intra-Uterine Device).
   * Additionally, male patients (including those who are vasectomized) whose partners are pregnant or might be pregnant must agree to use condoms for the duration of the treatment plan and for 90 days following completions of therapy.
   * Radiation therapy must have been completed at least 2 weeks prior to the enrollment date.
   * Patients with known brain metastases must have clinically controlled neurologic symptoms, defined as surgical excision and/or radiation therapy followed by 14 days of stable neurologic function prior to the first dose of study drug.
   * Ability to understand and the willingness to sign a written informed consent document.
2. Exclusion Criteria

   * Prior treatment with PARP inhibitor (excluding iniparib). Patients participating in protocol 7161 (NCI-2010-00356) are eligible.
   * Clinically significant and uncontrolled major medical condition(s) including but not limited to:
   * Active uncontrolled infection;
   * Symptomatic congestive heart failure;
   * Unstable angina pectoris or cardiac arrhythmia;
   * Psychiatric illness/social situation that would limit compliance with protocol requirements;
   * Any medical condition, which in the opinion of the investigator, places the patient at an unacceptably high risk for toxicities;
   * Myelodysplastic syndrome;
   * History of seizures within last 12 months or known neurological disorder pre-disposing to seizures
   * Patient is pregnant or lactating.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Cancer Care Allliance, Seattle, Washington, United States

REFERENCES:
- [Background] Chiarugi A. Poly(ADP-ribose) polymerase: killer or conspirator? The 'suicide hypothesis' revisited. Trends Pharmacol Sci. 2002 Mar;23(3):122-9. doi: 10.1016/S0165-6147(00)01902-7. PMID 11879679
- [Background] Virag L, Szabo C. The therapeutic potential of poly(ADP-ribose) polymerase inhibitors. Pharmacol Rev. 2002 Sep;54(3):375-429. doi: 10.1124/pr.54.3.375. PMID 12223530
- [Background] Sharpless NE, DePinho RA. Telomeres, stem cells, senescence, and cancer. J Clin Invest. 2004 Jan;113(2):160-8. doi: 10.1172/JCI20761. PMID 14722605
- [Background] Curtin NJ, Wang LZ, Yiakouvaki A, Kyle S, Arris CA, Canan-Koch S, Webber SE, Durkacz BW, Calvert HA, Hostomsky Z, Newell DR. Novel poly(ADP-ribose) polymerase-1 inhibitor, AG14361, restores sensitivity to temozolomide in mismatch repair-deficient cells. Clin Cancer Res. 2004 Feb 1;10(3):881-9. doi: 10.1158/1078-0432.ccr-1144-3. PMID 14871963
- [Background] Farmer H, McCabe N, Lord CJ, Tutt AN, Johnson DA, Richardson TB, Santarosa M, Dillon KJ, Hickson I, Knights C, Martin NM, Jackson SP, Smith GC, Ashworth A. Targeting the DNA repair defect in BRCA mutant cells as a therapeutic strategy. Nature. 2005 Apr 14;434(7035):917-21. doi: 10.1038/nature03445. PMID 15829967
- [Background] Bryant HE, Schultz N, Thomas HD, Parker KM, Flower D, Lopez E, Kyle S, Meuth M, Curtin NJ, Helleday T. Specific killing of BRCA2-deficient tumours with inhibitors of poly(ADP-ribose) polymerase. Nature. 2005 Apr 14;434(7035):913-7. doi: 10.1038/nature03443. PMID 15829966
- [Background] Wielckens K, Garbrecht M, Kittler M, Hilz H. ADP-ribosylation of nuclear proteins in normal lymphocytes and in low-grade malignant non-Hodgkin lymphoma cells. Eur J Biochem. 1980 Feb;104(1):279-87. doi: 10.1111/j.1432-1033.1980.tb04426.x. PMID 6245868
- [Background] Hirai K, Ueda K, Hayaishi O. Aberration of poly(adenosine diphosphate-ribose) metabolism in human colon adenomatous polyps and cancers. Cancer Res. 1983 Jul;43(7):3441-6. PMID 6406058